CLINICAL TRIAL: NCT01284517
Title: A Randomized, 6-week Double-blind, Placebo-controlled, Flexible-dose, Parallel-group Study of Lurasidone Adjunctive to Lithium or Divalproex for the Treatment of Bipolar I Depression in Subjects Demonstrating Non-response to Treatment With Lithium or Divalproex Alone.
Brief Title: Lurasidone HCI - A 6-week Phase 3 Study of Patients With Bipolar I Depression
Acronym: PREVAIL3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1050292; 2010-019778-34 (EudraCT Number)
Record Dates: First submitted 2011-01-25; First posted 2011-01-27 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-10

CONDITIONS: Bipolar Depression
Keywords: Bipolar I Depression; Lurasidone; Latuda
MeSH Terms: conditions — Bipolar Disorder | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lurasidone 20-120 mg flexible dose (Experimental)
  Interventions: Drug: Lurasidone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lurasidone — Tablets 20-120 mg, PM dosing,daily for 6 weeks
  Other Names: Latuda
  Arms: Lurasidone 20-120 mg flexible dose
Drug: Placebo — Equivalent to Lurasidone dosing
  Arms: Placebo

SUMMARY:
Lurasidone HCI is a compound that is a candidate for the treatment of bipolar I depression. This clinical study is designed to test the hypothesis that Lurasidone in combination with either Lithium or Divalproex is effective among patients with bipolar I depression.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent and is 18 to 75 years of age inclusive.
2. Meets DSM-IV-TR criteria for bipolar I disorder, most recent episode depressed (≥ 4 weeks and less than 12 months) without psychotic features.
3. Has a lifetime history of at least one bipolar manic or mixed manic episode.
4. Currently being treated with lithium or divalproex or willing to begin treatment with lithium or divalproex.
5. Not pregnant or nursing and is not planning pregnancy within the projected duration of the study.
6. Females of reproductive potential agree to remain abstinent or use adequate and reliable contraception throughout the study and for at least 30 days after
7. Good physical health on the basis of medical history, physical examination, and laboratory screening.

Exclusion Criteria:

1. Subject is considered by the investigator to be at imminent risk of suicide or injury to self, others, or property.
2. Any chronic organic disease of the CNS (other than Bipolar I Disorder).
3. Hospitalization for a manic or mixed episode within the past two months.
4. Used investigational compound within past 6 months.
5. Clinically significant history of alcohol or substance abuse within the past 3 months or alcohol or substance dependence within the past 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2010-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (75):
- United States (22):
  - Clinical Innovations, Inc., Costa Mesa, California
  - Clinical Innovations Inc., Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Clinical Innovations inc., Santa Ana, California
  - Collaborative Neuroscience Network, Torrance, California
  - Colorado Clinical Trials Inc., Highlands Ranch, Colorado
  - Accurate Clinical Trials, Kissimmee, Florida
  - Clinical Neuroscience Solutions Inc., Orlando, Florida
  - Northwest Behavioral Research Center, Roswell, Georgia
  - Institute for Behavioral Medicine LLC, Smyrna, Georgia
  - Precise Research Centers, Flowood, Mississippi
  - Village Clinical Research Inc., New York, New York
  - Medical & Behavioral Health Research, New York, New York
  - Zarzar Psychiatric Associates, PLLC, Raleigh, North Carolina
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - FutureSearch Clinical Trials, LP, Dallas, Texas
  - Pillar Clinical Research, Dallas, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Summit Research Network (Seattle) LLC, Seattle, Washington
- Canada (4):
  - Clinical Research Group Edmonton Inc, Edmonton, Alberta
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - Pierre-Janet Hospital, Gatineau, Quebec
  - Hopital Louis-H Lafontaine, Montreal, Quebec
- Colombia (4):
  - Centro de Investigaciones y Proyectos en Neurociencias CIPNA, Barranquilla
  - Centro de Investigacion y Atencion para la Salud Mental, Bogotá
  - CISNE - UIC Campo Abierto, Bogotá
  - Hospital Mental de Antioquia, Cali
- Czechia (4):
  - Psychiatricka ambulance, Brno-mesto
  - Vojenska nemocnice Olomouc, Olomouc
  - Clintrial, s.r.o., Prague
  - Psychiatry Trial s.r.o., Prague
- India (11):
  - Brain Mind Behavior Neuroscience Research Institute, Visakhapatnam, Andh Prad
  - Shanti Nursing Home, Kanchanpalli, Aurangabad, Maharashtra
  - SBKS Medical College and Hospital, Brij Psychiatry Hospital, Vadodara, Gujarat
  - Abhaya Hospital Psychiatry, Bangalore, Karna
  - K.S. Hegde Medical Academy, Mangalore, Karna
  - Poona Hospital & Research Center, Pune, Mahara
  - Mahatma Ghandi Institute of Medical Sciences, Wardha, Mahara
  - Mental Health Care & Research, Jaipur, Rajasthan
  - R.K. Yadav Memorial Mental Health & De-addiction Hospital, Jaipur, Rajasthan
  - Mahendru Psychiatric Center, Kanpur, Uttar Prad
  - Chatrapati Shau Maharaj Medical University, Lucknow, Utter Prad
- Japan (6):
  - Ongata Hospital, Hachioji-shi
  - Kohnodai Hospital, National Center for Global Health & Medicine, Ichikawa
  - National Hospital Organization Hizen Psychiatric Center, Kanzaki-gun
  - National Center of Neurology & Psychiatry, Kodaira-shi
  - Asakayama General Hospital, Sakaishi
  - Osaka Institute of Clinical Psychiatry Shin-abuyama Hospital, Takatsuki
- Lithuania (5):
  - Neuromeda JSC, Kaunas
  - Ziegzdriai Mental Hospital, Public Institution, Kaunas
  - Silutes Mental Health & Psychtherapy Center, JSC, Šilutė
  - Seskines Outpatient Clinic, Public Institution, Vilnius
  - Zirmunai Mental Health Center, Public Institution, Vilnius
- Peru (3):
  - Hospital Nacional Arzobispo Loayza, Lima
  - Hospital Nacional Hipolito Unanue, Lima
  - Clinica Vesalio, Lima
- Slovakia (8):
  - Centrum zdravia R. B. K. s.r.o., Bardejov
  - Bojniciach, Bojnice
  - Psychiatricka ambulancia Mentum s.r.o., Bratislava
  - FNsP Bratislava, Nemocnica Ruzinov, Bratislava
  - Nemocnica s poliklinikou Liptovsky Milulas, Liptovský Mikuláš
  - PsychoLine s.r.o., Rimavská Sobota
  - Nemocnica s poliklikou Sv. Barbory, Rožňava
  - Pro mente sana, Trenčín
- Ukraine (8):
  - Kherson Regional Psychiatric Hospital, Kherson, Vil Stepanivka
  - Dnipropetrovsk Regional Clinical Hospital named Mechnikov, Dnipropetrovsk
  - Com Inst Knipropetrovsk Reg Cl Psych Hospital DSMA, Dnipropetrovsk
  - St. In. Inst of Neurol, Psych, and Narcol of the AMSU, Kharkiv
  - Kyiv City Psychoneurological Hospital #2, Kyiv
  - Lviv Regional Clinical Psychiatric Hospital, Lviv
  - Ternopil Regional Municipal Dispensary, Narcology Dept., Ternopil
  - Zapor. Reg. CI Hospital, Zaporizhzhia SMU, Zaporizhzhya

REFERENCES:
- [Derived] Hopkins SC, Tomioka S, Szabo ST, Koblan KS. A clinical trial inclusion criteria to enrich for patients presenting with canonical symptom structure in bipolar depression. Contemp Clin Trials. 2024 Oct;145:107644. doi: 10.1016/j.cct.2024.107644. Epub 2024 Aug 3. PMID 39098761
- [Derived] Suppes T, Kroger H, Pikalov A, Loebel A. Lurasidone adjunctive with lithium or valproate for bipolar depression: A placebo-controlled trial utilizing prospective and retrospective enrolment cohorts. J Psychiatr Res. 2016 Jul;78:86-93. doi: 10.1016/j.jpsychires.2016.03.012. Epub 2016 Mar 31. PMID 27089521

RESULTS

PARTICIPANT FLOW:
Groups:
- Lurasidone 20-120 mg Flexible Dose+Li/VPA: Lurasidone 20-120 mg/day (PO) flexibly dosed+Lithium/divalproex
- Placebo + Li/VPA: Placebo + Lithium/divalproex
Period: Overall Study
Arm/Group | Lurasidone 20-120 mg Flexible Dose+Li/VPA | Placebo + Li/VPA
Started | 180 | 176
Completed | 148 | 140
Not Completed | 32 | 36

BASELINE CHARACTERISTICS:
Population: This is the full analysis set (intent-to-treat population)
Groups:
- Total: Total of all reporting groups
Arm/Group | Lurasidone 20-120 mg Flexible Dose+Li/VPA | Placebo + Li/VPA | Total
Number analyzed (Participants) | 176 | 166 | 342
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 0 | 3
  Between 18 and 65 years | 166 | 161 | 327
  >=65 years | 7 | 5 | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 43.1 (11.90) | 44.1 (11.99) | 43.6 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 93 | 184
  Male | 85 | 73 | 158
Region of Enrollment [Number; unit: participants]
  United States | 71 | 63 | 134
  Czech Republic | 9 | 8 | 17
  Slovakia | 17 | 21 | 38
  Canada | 9 | 8 | 17
  Ukraine | 17 | 14 | 31
  Lithuania | 10 | 9 | 19
  Peru | 6 | 7 | 13
  Colombia | 12 | 10 | 22
  Japan | 5 | 4 | 9
  India | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Endpoint (Week 6)
Description: MADRS total score ranges from a minimum of 0 to a maximum of 60. Lower values represent a better score, higher values represent a worse score. Similarly, greater negative change from baseline represents improvement, and positive changes from baseline represent worsening.
Time Frame: Baseline to week 6
Population: Full analysis set (intent-to-treat population)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo + Li/VPA: Placebo (PO) + Lithium or divalproex
Arm/Group | Lurasidone 20-120 mg Flexible Dose+Li/VPA | Placebo + Li/VPA
Number analyzed (Participants) | 176 | 166
units on a scale | -11.8 (0.76) | -10.4 (0.79)
Statistical Analysis 1: Comparison: Lurasidone 20-120 mg Flexible Dose+Li/VPA vs Placebo + Li/VPA; Null hypothesis (H0) assumes equal values between analysis groups in mean change from baseline in MADRS score, alternative hypothesis (HA) assumes unequal values between groups. Sample size determined by two-sample t-test. A mean difference of 3.25 units in change in MADRS score for the Lurasdone 20-120 mg arm over placebo with common standard deviation of 9 units was used. N=162 subjects per arm (total N=324) yields power of 90%. A 5% adjustment for drop-outs gives N=340, or N=170 per arm; Test type: Superiority or Other; p = 0.176, Mixed Models Analysis; Mean Difference (Final Values) = -1.5, Standard Error of Mean 1.08

2. Secondary Outcome: Mean Change From Baseline to Endpoint (Week 6) in: Clinical Global Impression Bipolar Version, Severity of Illness (CGI-BP-S) Score (Depression)
Description: CGI-EP-S depression score ranges from a minimum of 0 to a maximum of 7. Lower values represent a better score, higher values represent a worse score. Similarly, greater negative change from baseline represents improvement, and positive changes from baseline represent worsening.
Time Frame: Baseline to week 6
Population: Full analysis set (intent-to-treat population)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone 20-120 mg Flexible Dose+Li/VPA | Placebo + Li/VPA
Number analyzed (Participants) | 176 | 166
units on a scale | -1.36 (0.099) | -1.13 (0.102)
Statistical Analysis 1: Comparison: Lurasidone 20-120 mg Flexible Dose+Li/VPA vs Placebo + Li/VPA; Test type: Superiority or Other; p = 0.095, Mixed Models Analysis; Mean Difference (Final Values) = -0.24, Standard Error of Mean 0.141

3. Secondary Outcome: Mean Change From Baseline to Endpoint (Week 6) in: Sheehan Disability Scale (SDS) Total Score
Description: SDS total score ranges from a minimum of 0 to a maximum of 30. Lower values represent a better score, higher values represent a worse score. Similarly, greater negative change from baseline represents improvement, and positive changes from baseline represent worsening.
Time Frame: Baseline to week 6
Population: Full analysis set (intent-to-treat population)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone 20-120 mg Flexible Dose+Li/VPA | Placebo + Li/VPA
Number analyzed (Participants) | 176 | 166
units on a scale | -5.4 (0.85) | -5.4 (0.74)
Statistical Analysis 1: Comparison: Lurasidone 20-120 mg Flexible Dose+Li/VPA vs Placebo + Li/VPA; Test type: Superiority or Other; p = 0.992, ANCOVA; Mean Difference (Final Values) = 0.0, Standard Error of Mean 1.00

ADVERSE EVENTS:
Time Frame: 13 December 2010 to 7 August 2012
Description: Adverse event data (including number of participants at risk) is presented for the safety population, defined as subjects with exposure to at least one dose of study medication.
Groups:
- Placebo + Li/VPA: Placebo (PO)+ Lithium/divalproex
Arm/Group | Lurasidone 20-120 mg Flexible Dose+Li/VPA | Placebo + Li/VPA
Serious Adverse Events (participants affected / at risk) | 5/177 | 3/171
Other Adverse Events (participants affected / at risk) | 79/177 | 63/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 20-120 mg Flexible Dose+Li/VPA (N=177) | Placebo + Li/VPA (N=171)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Intentional Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaphylactic Shock (Immune system disorders) | 1 (1) | 0 (0)
Disease Progression (General disorders) | 1 (1) | 0 (0)
Depression Suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 20-120 mg Flexible Dose+Li/VPA (N=177) | Placebo + Li/VPA (N=171)
Akathisia (Nervous system disorders) | 25 (29) | 9 (12)
Nausea (Gastrointestinal disorders) | 18 (25) | 16 (20)
Headache (Nervous system disorders) | 15 (18) | 15 (16)
Insomnia (Psychiatric disorders) | 15 (16) | 18 (19)
Somnolence (Nervous system disorders) | 15 (16) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 14 (15) | 10 (13)
Tremor (Nervous system disorders) | 11 (14) | 9 (9)
Dizziness (Nervous system disorders) | 9 (9) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication; provided, if a multicenter publication is not forthcoming within 24 months following completion of study at all sites, the PI shall be free to publish.